CLINICAL TRIAL: NCT04930822
Title: Does Bioness Integrated Therapy System (BITS) Touch Screen Technology Improve Field Awareness to Inpatients With Neurological Visual Field Deficits
Brief Title: Evaluation of Bioness Integrated Therapy System (BITS) Touch Screen Technology to Improve Field Awareness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaylord Hospital, Inc (Other)
Collaborators: Connecticut Community Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202005FAG
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Neurologic Disorder; Traumatic Brain Injury; Acquired Brain Injury
Keywords: Visual Field Cut; Visual Field Interventions; Visual Field Impairments; Hemianopsia; Quadrantanopia; Long Term Acute Care Hospital; Occupational Therapy; Activities of Daily Living; Visual Neglect; Visual Inattention; Hemi-inattention; Touch Screen Technology; Visual Scanning
MeSH Terms: conditions — Stroke; Nervous System Diseases; Brain Injuries, Traumatic; Brain Injuries; Hemianopsia

STUDY DESIGN:
Intervention Model Description: Participants will be assigned into "A" and "B" groups upon admission in alternating fashion. The control group "A" will be prescribed conventional (table top, pen and paper) vision interventions provided by an occupational therapist and will receive pre- and post- assessment of visual field awareness. Treatment group "B" will include a prescribed regimen with use of BITS touch screen technology. Group B participants will receive the same pre- and post- assessment of visual field awareness as Group A participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Table Top Visual Intervention (Active Comparator): Interventions will include six, 20 minute sessions using pen and paper word search, scanning activities, and saccade visual training. All activities will be conducted with an occupational therapist/investigator.
  Interventions: Other: Table Top Visual Intervention
- Bioness Integrated Therapy System Visual Intervention (Experimental): Intervention will includes six sessions using the Bioness Integrated Therapy System for 20 minutes using the programs of visual scanning, visual pursuits and/or visual motor.All activities will be conducted with an occupational therapist/investigator.
  Interventions: Device: Bioness Integrated Therapy System Visual Intervention

INTERVENTIONS:
Other: Table Top Visual Intervention — Table top visual interventions and exercises.
  Other Names: Group A; Analog; Table Top
  Arms: Table Top Visual Intervention
Device: Bioness Integrated Therapy System Visual Intervention — Digital visual interventions and exercises.
  Other Names: Group B; Digital; BITS
  Arms: Bioness Integrated Therapy System Visual Intervention

SUMMARY:
The Bioness Integrated Therapy System (BITS) (Bioness Inc. Valencia, CA) Touch Screen is an FDA approved device comprised of an interactive touchscreen and diverse program options to challenge patients through the use of visual motor activities, visual and auditory processing, cognitive skills, and endurance training. The purpose of this study is to enroll a small group of adults currently undergoing inpatient rehabilitation, who were admitted for an acute neurological event and present with an acute neurological visual field impairment. The primary objective is to compare any increase in visual field awareness using a prescribed regimen consisting of conventional vision exercises compared with a regimen using BITS touch screen technology. Participants will be alternately assigned into "A" and "B" groups upon enrollment. The control group "A" will be prescribed conventional (table top, pen and paper) vision interventions provided by an occupational therapist and will receive pre- and post- assessment of visual field awareness. Treatment group "B" will include a prescribed regimen with use of BITS touch screen technology. Group B participants will receive the same pre- and post- assessment of visual field awareness as Group A participants. The hypothesis is that incorporation of the BITS touch screen technology, being more interactive, will result in better outcomes for visual field awareness. This is an unblinded quasi-randomized control trial that will determine best treatment intervention for visual field impairment. Safety will be measured by the number of reported adverse events. The study period will include 6 sessions per participant, conducted at one site, with the objective of enrolling at least 30 participants to have 15 participants in each study group.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the effectiveness of a multi-session prescribed regimen involving the Bioness Integrated Therapy System (BITS) touch screen technology as a safe, practical, and beneficial means to increase visual field awareness for individuals with neurological vision field deficits receiving inpatient therapy. The overall goal is to determine if the use of BITS touch screen technology more effectively improves visual field awareness than conventional vision interventions involving table-top pen and paper activities.

Prior to consenting interested individuals, the presence of a visual field deficit will be confirmed through confrontation testing. Consented participants will perform an initial Bells Test assessment to determine initial visual field awareness. In addition to the Bells Test assessment, a Neuro-Optometrist/investigator will use a Kinetic Field Analyzer to perform a visual field test to measure the density of the field deficit, or blind-spot. Bells Test and Kinetic Field Analyzer testing will be conducted within 1 week of admission to the study (pre-assessment) and within 1 week prior to participant discharge (post-assessment).

Consented participants will be alternately assigned to either Group "A" or Group "B". Participants in Group A will be offered traditional vision interventions that will include word search, scanning activities, and saccade training. Participants in Group B will be prescribed and complete a BITS regimen with occupational therapist/investigator using the BITS programs of visual scanning, visual pursuits and/or visual motor. Participants in both groups will complete six, 20 minute, sessions over three-weeks. A convenience sample of 30 participants (15 per group) will be recruited; the enrollment period is expected to last approximately 12 months.

In addition to the visual intervention, all participants will be evaluated by the Neuro-Optometrist/investigator for the need of prismatic correction for field expansion therapy. Prismatic correction is customarily used by eye care professionals to correct ocular deviations and align the eyes to correct double vision. This correction uses unequal prismatic correction for each eye. Prismatic correction can also be used in equal powers for each eye that is often called "yoked" prismatic correction. Yoked prisms are often used with stroke patients since they can change the location of objects in space as well as have the ability to balance visual skews in spatial perception. These patients often present with hemianopic visual field deficits. The yoked prism allows areas that are not seen to be perceived by displacing the objects into the area of vision not blinded by the stroke as well as balancing visual-spatial perceptual impairments. In turn this treatment allows rehabilitative therapy to be more effective with better outcomes and is part of the standard of care. All participants will be evaluated and receive the appropriate prismatic correction as prescribed.

Data analysis: All data will be collected and analyzed in an unpaired fashion as appropriate; adjustments for abnormal distribution, unequal variance, and repeated measure will be applied as necessary. In the case of missing or inconsistent data due to early withdraw, early participant discharge, or other unforeseen events, the datasets will be evaluated as normal.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years or older who are able to provide consent or have Power of Attorney (POA) able to consent.
* Must have an acute or subacute (diagnosed within the last 3 months) neurological diagnosis with a visual field deficit as verified by occupational therapist via confrontation testing.
* Admitted for inpatient rehabilitation
* Demonstrate the ability to follow 1 step directions
* Demonstrate sufficient upper extremity strength (as deemed appropriate by occupational therapist) to utilize BITS touch screen technology
* Ability to tolerate at least 30 minutes of intervention at a seated wheelchair level.

Exclusion Criteria:

* Severe cognitive impairments: Unable to follow one step directions, inability to communicate pain, or to stop intervention if needed
* Quadriparesis
* Previous significant visual impairment impacting visual fields or resulting in legal blindness in past medical history
* Re-admitted to Acute Care and do not return within 1 week
* Currently on a ventilator for respiratory support
* Unstable vital signs or deemed inappropriate to participate in therapy per Medical Staff
* Uncontrolled or new (within 24 hours) arrhythmias.
* Unresolved or new (within 24 hours) deep vein thrombosis.
* Concurrent severe neurological pathology/disease or stroke within 72 hours.
* Any reason the physician may deem as harmful to the participant to enroll or continue in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Fagan, OTR/L, Principal Investigator — Gaylord Specialty Healthcare
Locations (1):
- Gaylord Hospital, Wallingford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Copies of the study protocol will be provided upon request. Requests for copies of the de-identified research data will be considered on a situational basis.

REFERENCES:
- [Background] Master CL, Scheiman M, Gallaway M, Goodman A, Robinson RL, Master SR, Grady MF. Vision Diagnoses Are Common After Concussion in Adolescents. Clin Pediatr (Phila). 2016 Mar;55(3):260-7. doi: 10.1177/0009922815594367. Epub 2015 Jul 7. PMID 26156977
- [Background] Sara Stephenson, Alice Anderson-Tome, Sarah Fischer, Abby Guzman, William Meredith, Chandler Somers; Pilot Study: Using the Bioness Integrated Therapy System (BITS) To Examine the Correlation Between Skills and Success With On-the-Road Driving Evaluations. Am J Occup Ther 2019;73(4_Supplement_1):7311515280. https://doi.org/10.5014/ajot.2019.73S1-PO4054
- [Background] Goodwin D. Homonymous hemianopia: challenges and solutions. Clin Ophthalmol. 2014 Sep 22;8:1919-27. doi: 10.2147/OPTH.S59452. eCollection 2014. PMID 25284978
- [Background] Gauthier L, Dehaut F, Joanette Y. The Bells Test: A quantitative and qualitative test for visual neglect. International Journal of Clinical Neuropsychology. US: MelNic Press, Inc.; 1989;11(2):49-54.
- See also: Britannica. Visual Field Defect — https://www.britannica.com/science/visual-field-defect
- See also: Visual Field Testing. Cleveland Clinic — https://my.clevelandclinic.org/health/diagnostics/14420-visual-field-testing
- See also: Visual Field Testing. American Academy of Ophthalmology — https://www.aao.org/eye-health/tips-prevention/visual-field-testing

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Table Top Visual Intervention | Bioness Integrated Therapy System Visual Intervention
Started | 18 | 19
Completed | 16 | 17
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Table Top Visual Intervention | Bioness Integrated Therapy System Visual Intervention | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (18.4) | 63.4 (13.6) | 63.2 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Bells Test
Description: Used to determine initial visual field awareness. The participant is presented with a standardized pen and paper assessment that includes pictures of bells and other objects. The participant has to locate and circle as many bells as they can without circling any distractors. The participant is scored on the time that it takes to complete the assessment, the number of bells that are located on both the left and right side of the page, and the number of distractors that are located. The Bells test scored on a scale of 0 through 35; the higher the score the better.
Time Frame: Pre and post tests will be collected within 1 week following enrollment and within 1 week prior to discharge, approximately 1 month from baseline.
Population: Number of total items correct
Measure: Mean (95% Confidence Interval); unit: Number of items correct
Groups:
- Pre-Assessment Tabletop; Pre-Assessment BITS: Bells test score prior to intervention
- Post-Assessment Tabletop; Post-Assessment BITS: Bells test score post intervention
Arm/Group | Pre-Assessment Tabletop | Post-Assessment Tabletop | Pre-Assessment BITS | Post-Assessment BITS
Number analyzed (Participants) | 16 | 16 | 17 | 17
Number of items correct | 14.2 [8.0 to 20.4] | 18.3 [12.8 to 23.7] | 19.3 [13.2 to 25.4] | 27.1 [22.4 to 31.7]
Statistical Analysis 1: Comparison: Pre-Assessment Tabletop vs Pre-Assessment BITS; Alpha set at 0.05; Test type: Superiority; p = 0.1779, ANOVA — Fisher's LSD utilized; no correction for multiple comparisons; Predicted least squares mean difference = -5.107, 95% CI 2-sided [-12.60 to 2.385]
Statistical Analysis 2: Comparison: Post-Assessment Tabletop vs Post-Assessment BITS; Alpha set at 0.05; Test type: Superiority; p = 0.0219, ANOVA — Fisher's LSD utilized; no corrections for multiple comparisons; Predicted least squares mean difference = -8.809, 95% CI 2-sided [-16.30 to -1.317]
Statistical Analysis 3: Comparison: Pre-Assessment Tabletop vs Post-Assessment Tabletop; Alpha set at 0.05; Test type: Superiority; p = 0.0139, ANOVA — Fisher's LSD utilized; no corrections for multiple comparisons; Predicted least squares mean difference = -4.063, 95% CI 2-sided [-7.240 to -0.8849]
Statistical Analysis 4: Comparison: Pre-Assessment BITS vs Post-Assessment BITS; Alpha set at 0.05; Test type: Superiority; p < 0.0001, ANOVA — Fisher's LSD utilized; no corrections for multiple comparisons; Predicted least squares mean difference = -7.765, 95% CI 2-sided [-10.85 to -4.682]

2. Primary Outcome: Kinetic Field Assessment - Field of View
Description: Neuro-Optometrist delivered test. Measures the density or presence of field deficits, or blind-spots, in participants using moving objects with a fixed luminance and color. Each participant has both eyes assessed (n = 2). Measured in degrees from 0-360, typical values for healthy adults are 170-200 degrees.
Time Frame: Pre and post tests will be collected within 1 week following enrollment and within 1 week prior to discharge.
Population: Total Field of View
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Eyes
Groups:
- Pre-Exam Tabletop; Pre-Exam BITS: Pre intervention kinetic field test administered by a neuro-optometrist.
- Post-Exam Tabletop; Post-Exam BITS: Post intervention kinetic field test administered by a neuro-optometrist.
Arm/Group | Pre-Exam Tabletop | Post-Exam Tabletop | Pre-Exam BITS | Post-Exam BITS
Number analyzed (Participants) | 13 | 13 | 16 | 16
Number analyzed (Eyes) | 25 | 25 | 32 | 32
Degrees | 117.68 (43.68) | 167 (49.38) | 125.56 (44.36) | 180.97 (34.78)
Statistical Analysis 1: Comparison: Pre-Exam Tabletop vs Pre-Exam BITS; Alpha set at 0.05; Test type: Superiority; p = 0.4930, ANOVA — Fisher's LSD utilized; no correction for multiple comparisons; Predicted least squares mean difference = -7.883, 95% CI 2-sided [-30.59 to 14.83]
Statistical Analysis 2: Comparison: Post-Exam Tabletop vs Post-Exam BITS; Alpha set at 0.05; Test type: Superiority; p = 0.2255, ANOVA — Fisher's LSD utilized; no correction for multiple comparisons; Predicted least squares mean difference = -13.97, 95% CI 2-sided [-36.68 to 8.744]
Statistical Analysis 3: Comparison: Pre-Exam Tabletop vs Post-Exam Tabletop; Alpha set at 0.05; Test type: Superiority; p < 0.0001, ANOVA — Fisher's LSD utilized; no correction for multiple comparisons; Predicted least squares mean difference = -49.32, 95% CI 2-sided [-63.18 to -35.46]
Statistical Analysis 4: Comparison: Pre-Exam BITS vs Post-Exam BITS; Alpha set at 0.05; Test type: Superiority; p < 0.0001, ANOVA — Fisher's LSD utilized; no correction for multiple comparisons; Predicted least squares mean difference = -55.41, 95% CI 2-sided [-67.66 to -43.16]

3. Primary Outcome: Kinetic Field Testing - Visual Field Index
Description: Neuro-Optometrist delivered test. Measures the density or presence of field deficits, or blind-spots, in participants using moving objects with a fixed luminance and color. Each participant has both eyes assessed (n = 2). Visual Field Index is a percentage from 0-100%, with 100% being a normal field and 0% being a perimetrically blind field.
Time Frame: Pre and post tests will be collected within 1 week following enrollment and within 1 week prior to discharge.
Population: Visual Field Index = [(Kinetic field measurement) / (normative value)] * 100
Measure: Mean (Standard Deviation); unit: Visual field index
Units Other Than Participants: Eyes
Arm/Group | Pre-Exam Tabletop | Post-Exam Tabletop | Pre-Exam BITS | Post-Exam BITS
Number analyzed (Participants) | 13 | 13 | 16 | 16
Number analyzed (Eyes) | 25 | 25 | 32 | 32
Visual field index | 38.96 (14.46) | 55.29 (16.35) | 41.58 (14.69) | 59.92 (11.52)
Statistical Analysis 1: Comparison: Pre-Exam Tabletop vs Pre-Exam BITS; Alpha is set at 0.05; Test type: Superiority; p = 0.49, ANOVA — Fisher's LSD utilized; no correction for multiple comparisons; Predicted least squares mean difference = -2.611, 95% CI 2-sided [-10.13 to 4.909]
Statistical Analysis 2: Comparison: Post-Exam Tabletop vs Post-Exam BITS; Alpha set at 0.05; Test type: Superiority; p = 0.2246, ANOVA — Fisher's LSD utlilized; no correction for multiple comparisons; Predicted least squares mean difference = -4.634, 95% CI 2-sided [-12.15 to 2.886]
Statistical Analysis 3: Comparison: Pre-Exam Tabletop vs Post-Exam Tabletop; Alpha set at 0.05; Test type: Superiority; p < 0.0001, ANOVA — Fisher's LSD; no correction for multiple comparisons; Predicted least squares mean difference = -16.32, 95% CI 2-sided [-20.91 to -11.74]
Statistical Analysis 4: Comparison: Pre-Exam BITS vs Post-Exam BITS; Alpha set at 0.05; Test type: Superiority; p < 0.0001, ANOVA — Fisher's LSD utilized; no correction for multiple comparisons; Predicted least squares mean difference = -18.35, 95% CI 2-sided [-22.40 to -14.29]

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events during the course of enrollment in study activities, approximately 1 month from baseline to hospital discharge.
Arm/Group | Table Top Visual Intervention | Bioness Integrated Therapy System Visual Intervention
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT04930822/Prot_SAP_000.pdf